CLINICAL TRIAL: NCT00173940
Title: Collection of Blood and Urine Specimens From Volunteers Utilizing Health Examination Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100203282
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2002-07

CONDITIONS: Chronic Diseases; Hypertension; Diabetes; Obesity; Chronic Renal Failure
Keywords: chronic diseases, such as hypertension, diabetes, obesity, chronic renal failure, and so on
MeSH Terms: conditions — Chronic Disease; Hypertension; Diabetes Mellitus; Obesity; Kidney Failure, Chronic

SUMMARY:
In summary, the researchers want to construct a longitudinal data bank using voluntary health examination participants. Researchers in the National Taiwan University Hospital (NTUH) campus can utilize these data to clarify the effects of several genetic and environmental factors on various common diseases in Taiwan in the future.

ELIGIBILITY:
Inclusion Criteria:

* Persons who sign informed consent

Exclusion Criteria:

* Age below 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Jen Yen, MD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan